

## **Main Study Information Letter**

**Title of Study:** Supporting Parents to Choose Wisely: A Multi-Method Study to Increase Knowledge and Manage Expectations for Common Acute Childhood Conditions

# **Principal Investigator**

Lisa Hartling, PhD

Professor, Department of Pediatrics, Faculty of Medicine and Dentistry

University of Alberta, Edmonton, Alberta, Canada

Email: hartling@ualberta.ca Telephone: 780-492-6124

## **Co-Investigator**

Shannon Scott, PhD Professor, Faculty of Nursing

University of Alberta, Edmonton, Alberta, Canada

Email: shannon.scott@ualberta.ca

Telephone: 780-492-1037

Sarah Elliott, PhD

Department of Pediatrics, Faculty of Medicine and Dentistry

University of Alberta, Edmonton, Alberta, Canada

Email: se2@ualberta.ca Telephone: (780) 492-1241

### **Project Coordinator:**

Samantha Cyrkot, MSc

Department of Pediatrics, Faculty of Medicine and Dentistry

University of Alberta, Edmonton, Alberta, Canada

Email: archecho@ualberta.ca Telephone: (780) 492-1241

You are being invited to take part in an online research study. Before you agree to take part, you can email the Project Coordinator, Samantha at <archecho@ualberta.ca> if you would like more information about this study. You are free to ask any questions about anything you do not understand. You will be able to download a copy of this letter for your records.

Why am I being asked to take part in this research study? You are being asked to take part in this study because you are over 18 years of age and the parent or legal guardian of a child under 5 years. You have either a computer, tablet or smartphone. You also have access to the Internet, email and know English. Parents living in Canada can participate.

What is the reason for doing the study? The reason for doing this study is to help parents increase their knowledge and manage expectations for common acute childhood conditions such as an ear



infection or a common cold. We have made six different blogshots. A blogshot is an image summarizing information. Each blogshot gives helpful information about a specific common acute childhood condition based on the advice from Choosing Wisely Canada. We are looking to see if these blogshots are easy to understand, helpful and useful for parents.

What will I be asked to do? You will randomly be assigned to Group A or Group B in this study. Group A will receive three of six blogshots over a 4-week period (a different blogshot will be sent by email to you each week for three weeks, then in the final week you will receive the same three blogshots in one summary email to review). Group B will receive the other three of six blogshots, following the same email sequence and timing. All participants from both groups will be asked to complete one baseline questionnaire at the start of the study and a follow-up questionnaire at week 5, month 3 and month 6 about different common acute childhood conditions, the blogshots and their content. The reason for assigning you into a group is to help us evenly share the blogshots between all participants. You will not be asked to interact with other members from your group or know who else has been assigned to the same group as you.

Nooro, an independent online survey company, has been selected to manage the database of survey responses on behalf of the University of Alberta. Nooro is compliant with the Personal Information Protection and Electronic Documents Act (PIPEDA), which took full effect on January 1st, 2004. They will be sending you automated email messages with links to the blogshots and questionnaires. Each blogshot will take about **5 minutes** to read. Each questionnaire will take about **15-20 minutes** to complete.

Below is a list of the study tasks that you will be asked to complete:

| Week 0 | Complete the baseline and demographic questionnaire. |
|---|---|
| Week 1 | Read one blogshot on a topic related to common acute childhood conditions. |
| Week 2 | Read one blogshot on a different topic related to common acute childhood conditions. |
| Week 3 | Read one blogshot on a different topic related to common acute childhood conditions. |
| Week 4 | Review all three blogshots from week 1-3. |
| Week 5 | Complete the first follow-up questionnaire and a 30-60 minute interview (optional). |
| Month 3 | Complete the second follow-up questionnaire. |
| Month 6 | Complete the third follow-up questionnaire. |

When you complete the week 5 follow-up questionnaire, you will be asked at the end if you would like to participate in a one-on-one interview with the Project Coordinator, Samantha. If you are interested, you will be interviewed to give your thoughts on the blogshots and your experience in this study. This interview will take 30-60 minutes. You will be contacted by email to schedule the online interview via Zoom video conferencing. You do not have to participate in the interview portion of the study if you do not want to. This is optional and will not affect the care that you or your child receive.

What are the risks and discomforts? This is a low risk study. This study will use Nooro to manage the study and collect data. This is an externally hosted service. While the Research Ethics Board of the University of Alberta has approved using Nooro to collect data for this study, there is a small risk of a privacy breach for data collected on external servers. If you are worried about



this, we would be happy to make other plans such as doing the questionnaires by telephone. Please email Samantha at <a href="archecho@ualberta.ca">archecho@ualberta.ca</a> if you have any concerns. It is not possible to know all the risks that may happen in a study, but researchers have taken all reasonable safeguards to minimize any known risks to a study participant.

What are the benefits to me? There are no direct benefits to being in this study. But after viewing the blogshots, you will learn how to manage different conditions such as an ear infection or a common cold. There is also scientific benefit because the information you share through the questionnaires will be important for understanding how useful these blogshots are at sharing scientific information to parents in a user-friendly format.

**Do I have to take part in the study?** Being in this study is your choice. If you do decide to be in the study, you can change your mind and stop being in the study at any time. You can also stop being in the study at any point while completing the questionnaires or reviewing the blogshots by closing your web browser. You do not have to answer any questions that you do not want to answer. You can also stop being in the study by emailing Samantha at <a href="mailto:archecho@ualberta.ca">archecho@ualberta.ca</a> or contacting Dr. Elliott at <a href="mailto:se2@ualberta.ca">se2@ualberta.ca</a> or 780 492-1241.

After you submit a completed questionnaire or close your web browser (with partial responses entered), you will not be able to withdraw any data that you entered as it will become part of the data set.

Will I be paid to be in this research? To thank you for your time, you will receive a \$10 CAD electronic gift card for each follow-up questionnaire that you complete (to a maximum of \$30 CAD). If you choose to participate in the optional interview portion of the study, you will receive an additional \$25 CAD electronic gift card for your time.

Will my information be kept private? During this study we will do everything we can to make sure that all information you provide is kept private. No information relating to this study that includes your email will be released outside of the researcher's office or published by the researchers unless you give us your express permission. The study will not ask you any identifiable information beyond your first name and email address which will be separated from the main data set. Sometimes, by law, we may have to release your information with your name so we cannot guarantee absolute privacy. However, we will make every legal effort to make sure that your information is kept private. During research studies, it is also important that the data we get is accurate. For this reason, your data, including your name, may be looked at by people from the Research Ethics Board.

During the study, we will keep all electronic documents at the University of Alberta on secure servers with passwords. The only people who can see the data is the study team at the University of Alberta. After the study is done, we will still need to securely store your data that was collected as part of the study. However, your first name and email will be deleted after the study is done. We will keep all other electronic research documents secured for five years at the University of Alberta on secure servers with passwords. We will destroy the documents after five years. No paper copies will be stored. The information we get for this study may be looked at again in the



future to help us answer other study questions. If so, the ethics board will first review the study to ensure the information is used ethically.

Will I get a copy of the study findings? A summary of the study findings will be shared with you by email after the study is completed.

**What if I have questions?** If you have any questions about the research now or later, please email Samantha at <archecho@ualberta.ca> or Dr. Elliott at <se2@ualberta.ca>, or call 780 492-1241.

The plan for this study has been reviewed by a Research Ethics Board at the University of Alberta. If you have any questions regarding your rights as a research participant or how the research is being conducted you may contact the University of Alberta Research Ethics Office at <<u>reoffice@ualberta.ca</u>> or 780-492-2615 and quote Ethics ID Pro00116449. This office is independent of the study investigators.

This study has been funded by the Women and Children's Health Research Institute (WCHRI).

#### **Consent Statement**

I have read the above and consent to participate in this research study. I will receive a copy of this Study Information Letter for my records.

Please click here to download a copy of this Study Information Letter for your reference & records.

### I AGREE TO PARTICIPATE

By clicking this box, you indicate that you have read the information above and agree to participate in the study.